CLINICAL TRIAL: NCT07136402
Title: Massachusetts Community Engaged Alliance (MA-CEAL) Community Health Ambassador Program
Brief Title: MA-CEAL Community Health Ambassador Program
Acronym: CHANGE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn for study design changes prior to implementation of the study. No participants were enrolled.
Sponsor: Boston Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Massachusetts Community Engaged Alliance (MA-CEAL) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-45218; OT2HL158287 (NIH)
Record Dates: First submitted 2025-05-13; First posted 2025-08-22 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Hypertension; Diabetes Mellitus; Health Care Utilization
Keywords: Community health ambassadors (CHA); Community health centers; Workshops
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Patient Acceptance of Health Care

STUDY DESIGN:
Intervention Model Description: A waitlist-control trial design will be used for this study. 6 of the 12 participating housing developments will be randomized into the intervention arm and 6 into the control arm. At month 0 all participants will participate in baseline activities (surveys). At month 18 the control arm will begin the intervention. The whole study is projected to take 36 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Phase A) (Experimental): Community health centers randomized into this arm will receive study interventions in the first 18 months of the study.
  Interventions: Other: Educating participants about healthcare resources; Other: Healthcare appointments; Other: Workshops
- Control (Phase B) (Experimental): Community health centers randomized into this arm will be wait listed and will not receive study interventions during the first 18 months of the study. They will receive study interventions during the last 12 months of the study.
  Interventions: Other: Educating participants about healthcare resources; Other: Healthcare appointments; Other: Workshops

INTERVENTIONS:
Other: Educating participants about healthcare resources — MA-CEAL team members, including the community health ambassador (CHA), will assist in connecting residents with healthcare resources.
Other: Healthcare appointments — MA-CEAL team members, including the community health ambassador (CHA), will assist residents in making physician appointments.
Other: Workshops — Trained CHAs will provide workshops with information about diabetes and hypertension and how to be screened and get care.

SUMMARY:
This research is being conducted to investigate how to increase primary care health care visits and screenings and treatment for hypertension and diabetes in residents of housing developments in Boston. The investigators are partnering with Boston Housing Authority (BHA) and Trinity housing management to randomize 12 housing developments (6 in intervention and 6 in control). 6 residents from the housing developments will become Community Health Ambassadors (CHA). The CHAs will be trained to conduct "workshops" within the intervention arm. These workshops will cover Diabetes Mellitus (DM) and Hypertension (HTN) information. Along with the workshops, CHAs will act as mentors for the residents and provide them with resources to connect them to primary care, Community Health Centers, food pantry resources, how to get insurance, and other needed services. CHAs will be part-time employees of the Massachusetts Community Engaged Alliance (MA-CEAL), so they will be paid for the work they are doing while simultaneously building their professional skill set.

MA-CEAL's community engagement (CE) team will act as liaisons and mentors for the CHA's to help guide them and also connect them to opportunities for career/personal development.

ELIGIBILITY:
Inclusion Criteria:

* Current resident in selected Boston Health Authority (BHA) and Trinity housing developments
* Speak and understand English and/or Spanish

Exclusion Criteria:

* Does not speak English or Spanish
* Not a resident of the development

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Number of primary care visits | Baseline, 6 months, 12 months, 18 months
  Self-report primary care visits in the last 18 months will be obtained using selected items from the National Health Interview Survey (NHIS)

SECONDARY OUTCOMES:
Number of screenings for diabetes | Baseline, 6 months, 12 months, 18 months
  Self-reported by participants in a study questionnaire
Number of screenings for hypertension | Baseline, 6 months, 12 months, 18 months
  Self-reported by participants in a study questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Linas, MD MPH, Principal Investigator — Boston Medical Center, Infectious Disease

IPD SHARING:
Plan to Share IPD: No